CLINICAL TRIAL: NCT05975229
Title: The Effects of an 8-week Knitting Program on Osteoarthritis Symptoms in Elderly Women: A Pilot Randomized Controlled Trial
Brief Title: The Effects of a Knitting Program on Osteoarthritis Symptoms in Elderly Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Principal Investigator, Guillaume Léonard, Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H02-16-12
Record Dates: First submitted 2023-07-24; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis
Keywords: hand; osteoarthritis; exercise; knitting; women; pain; stiffness
MeSH Terms: conditions — Osteoarthritis; Motor Activity; Pain | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Single-blind, two-arm pilot RCT with a parallel group design
Who Masked: Outcomes Assessor
Masking Description: The trained independent evaluator conducting the performance evaluations and calculating the scores of the self-reported questionnaires was blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): Educational pamphlet and knitting program
  Interventions: Other: Knitting and education (pamphlet)
- control (Other): Educational pamphlet and assigned to a waiting list
  Interventions: Other: Education (pamphlet)

INTERVENTIONS:
Other: Knitting and education (pamphlet) — Pamphlet and knitting program (-8-week duration). The knitting program has two components: bi-weekly 20-minute group knitting sessions and 20-minute home daily knitting on the 5 remaining weekdays.
  Arms: experimental
Other: Education (pamphlet) — Receive only the pamphlet, not the knitting program.
  Arms: control

SUMMARY:
This pilot randomized controlled trial (RCT) studies the adherence and clinical effectiveness of a knitting program in older females suffering from hand osteoarthritis (HOA) to evaluate the acceptability of this intervention and assess the feasibility of a larger-scale RCT.

It is a single-blind, two-arm pilot RCT with a parallel group design with 40 participants (20 control, 20 experimental). Control participants are given an educational pamphlet and assigned to a waiting list. The knitting program (-8-week duration) has two components: bi-weekly 20-minute group knitting sessions and 20-minute home daily knitting on the 5 remaining weekdays. Measures include knitting adherence (implementation outcomes) as well as stiffness, pain, functional status, hand physical activity level, patient's global impression of change, health-related quality of life, self-efficacy, and grip strength (clinical outcomes measured throughout the 8-week program and 4 weeks after the intervention).

DETAILED DESCRIPTION:
Background: Exercise therapy is effective in reducing symptoms and disability associated with hand osteoarthritis (HOA) but has low adherence. An intervention consisting in a meaningful occupation, such as knitting, may improve adherence to treatment. This pilot randomized controlled trial (RCT) studies the adherence and clinical effectiveness of a knitting program in older females suffering from HOA to evaluate the acceptability of this intervention and assess the feasibility of a larger-scale RCT.

Methods: Single-blind, two-arm pilot RCT with a parallel group design with 40 participants (20 control, 20 experimental). Control participants are given an educational pamphlet and assigned to a waiting list. The knitting program (-8-week duration) has two components: bi-weekly 20-minute group knitting sessions and 20-minute home daily knitting on the 5 remaining weekdays. Measures included knitting adherence (implementation outcomes) as well as stiffness, pain, functional status, hand physical activity level, patient's global impression of change, health-related quality of life, self-efficacy, and grip strength (clinical outcomes measured throughout the 8-week program and 4 weeks after the intervention).

ELIGIBILITY:
Inclusion Criteria:

* Meet the clinical and radiographic criteria of definite HOA set out by the American College of Rheumatology (ACR) and have experienced pain symptoms for at least 3 months;
* Be a woman aged between 50 and 85 years; 3) have moderate to severe morning stiffness (defined as a score ≥ 4 on a 10 cm visual analogue scale at the time of study entry;
* Display X-ray evidence of joint space narrowing of the hands;
* Have no previous experience with knitting or have not knitted in the last 6 months;
* Be available for sessions at the senior's club twice weekly;
* Be able to understand written and verbal English instructions.

Exclusion Criteria:

* Suffered from other orthopedic or rheumatologic diseases (e.g., inflammatory arthritis), or showed evidence of chondrocalcinosis;
* Had a history of finger joint surgery;
* Suffered from an acute disease, such as uncontrolled diabetes mellitus, untreated hypertension, neurological deficits (motor or sensory), cognitive deficit or mental health conditions;
* Were taking OA medication that was expected to change during the study period;
* Were receiving current rehabilitation treatments or any other pain-related treatment besides medication for OA;
* Had received a corticosteroid injection in a finger joint within the last 6 months;
* Planned to move outside the region within 6 months.

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 37 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Stiffness | daily for 12 weeks
  0-100 visual analog scale where 0 = no stiffness, 100 = worst imaginable stiffness

SECONDARY OUTCOMES:
Dropout rates | week 8
  Assessed through a in-house questionnaire
Adherence to the knitting program | Baseline, week 4, week 8, and week 12
  It was estimated using the logbook and the seniors club attendance sheet, whereby we divided the number of knitting sessions completed (at the club and at home) by the number of knitting sessions prescribed (56 sessions)
pain level | Multiple times daily for 12 weeks
  0-100 visual analog scale where 0 = no pain, 100 = worst imaginable pain
Functional status | Baseline, week 4, week 8, and week 12
  Was assessed using the Australian/Canadian Osteoarthritis Hand Index (AUSCAN). It consists in a 15-item scale, with items grouped into three subsections: A) pain intensity, B) stiffness severity, and C) hand functional status/difficulty in activities of daily living. For each item, scores range from 0 (no symptoms) to 4 (severe symptoms)
Hand physical activity | Baseline, week 4, week 8, and week 12
  was measured using an adapted version of the 7-Day Physical Activity Readiness (PAR). It is in the form of a calendar in which participants record the duration (minutes per day) and frequency (days per week) of physical activity.
Patient's global impression of change | Baseline, week 4, week 8, and week 12
  It was assessed by asking patients if, following the knitting program, their condition was: 1) very much improved; 2) much improved; 3) minimally improved; 4) no change; 5) minimally worse; 6) much worse; 7) very much worse
Health-related Quality of life (QoL) | Baseline, week 4, week 8, and week 12
  It was evaluated using the EuroQoL Index (EQ-5D-5L), which covers mobility, self-care, daily activities, Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Self-efficacy | Baseline, week 4, week 8, and week 12
  It was assessed using The Stanford Arthritis Self-Efficacy Scale, consisting in statements which patients rate on a ten-point scale ranging from 1 (very uncertain) to 10 (very certain).
Bilateral hand grip strength | Baseline, week 4, week 8, and week 12
  It was measured using a portable JAMAR Hydraulic Hand Dynamometer in the standardized sitting position

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa, Ottawa, Quebec, Canada